CLINICAL TRIAL: NCT01785485
Title: IMPACT: Integrative Medicine PrimAry Care Trial: A Comparative Effectiveness Study of an Integrative Primary Care Clinic
Brief Title: IMPACT - Integrative Medicine PrimAry Care Trial
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Sally Dodds, Associate Professor/Research Scholar of Medicine & Psychiatry, University of Arizona
Other Study IDs: Coors001
Record Dates: First submitted 2013-01-31; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Adult Primary Care Patients
Keywords: Integrative medicine; primary care; cost-effectiveness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary care patients: Primary care patients who are members of UAIHC.
  Interventions: Other: Integrative medicine primary care model

INTERVENTIONS:
Other: Integrative medicine primary care model — An integrative medicine primary medical care as defined by the Arizona Center for Integrative Medicine.

SUMMARY:
This study is Phase II of a project by the University of Arizona Center for Integrative Medicine (AzCIM). Collaborating with AzCIM is the Health Outcomes and Pharmacoeconomics (HOPE) Center and the RAND Corporation, Inc. Phase II is a prospective evaluation of the clinical and cost effectiveness (outcomes) of an integrative medicine professional practice model for adult primary care delivery (the University of Arizona Integrative Health Center - UAIHC in Phoenix, AZ). Data will be gathered from eligible and consenting members of UAIHC. In addition, a fidelity evaluation will assess whether the practice model was implemented as planned.

The specific aims are to: 1) Recruit, consent, and enroll a sample of eligible patient and staff participants from UAIHC; 2) Conduct outcome evaluation of UAIHC care using patient data from medical records abstractions, self-report assessments, clinic administrative and service utilization/encounter data, and health insurance claims data; and, 3) Conduct fidelity evaluation of the implementation of the UAIHC model as described in its business plan using patient- and staff-reported fidelity assessments, random chart audits, and abstracted clinic administrative data.

Participants. 1) Participants from the clinic patient population for whom clinical and cost outcomes will be tracked (n=500); 2) Clinic patients from whom fidelity data will be collected (n=180); and, 3) Clinic personnel from whom fidelity data will also be collected (n=14).

Data Collection. For outcomes evaluation, data will be collected at baseline (initial clinic visit), and at 3-, 6-, and 12-month follow up periods. Sources include clinical symptoms and biomarkers from medical records abstractions; patient reported outcomes and satisfaction questionnaires; clinic service encounter logs; and, cost data from health insurance claims information and clinic financial data. For fidelity evaluation, data will be collected monthly for 6 months after study start, quarterly for the next 6 months, and semi-annually from then on. Patient data for fidelity will be gathered on a single randomized day of the week using a self-administered patient feedback questionnaire. For personnel, fidelity data will be collected at the same intervals using a self-administered provider perceptions questionnaire of inter-professional team and integrative medical care. Data from audits of randomly selected patient charts and administrative records will also be used.

ELIGIBILITY:
Outcomes Study Sample:

Inclusion Criteria:

* Enrollment in primary care (members) at UAIHC;
* Adults age 18 or older.

Exclusion Criteria:

* Currently pregnant at time of recruitment;
* Patients who attend the UAIHC clinic as consultation-only patients;
* Significant cognitive impairment to the extent that the individual is unable to understand consent and respond to questionnaires.

Fidelity Study Sample (Patients):

Inclusion Criteria:

* Enrollment in primary care (members) at UAIHC;
* Adults age 18 or older.

Exclusion Criteria:

* Significant cognitive impairment to the extent that the individual is unable to understand consent and respond to questionnaires.

Fidelity Study Sample (Providers):

Inclusion Criteria:

* All clinical and support personnel.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only patients who are enrolled in primary care (members) at UAIHC and who meet the inclusion/exclusion criteria are eligible to enroll in this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Total healthcare costs from the payer's perspective-total paid costs according to claims data. | 12 months of paid costs pre and post beginning membership at UAIHC

SECONDARY OUTCOMES:
1. Self-report instruments | Baseline, 3-, 6-, and 12-months
  Composite:
  Short Form -12 (Ware, 1996) WHO-5 Well-being Index (Bech, 2003) Perceived Stress Scale (Cohen 1983). Work Productivity and Activity Impairment (Reilly, 1993). Patient Activation Measure (Hibbard, 2004). Diet quality. Behavioral Risk Factor Surveillance System Fruits/Vegetables (CDC, 2012).
  Physical Activity. Behavioral Risk Factor Surveillance System Physical Activity (CDC, 2012).
  Stress burden (Littman, 2006). Depression. PHQ-2 (Kroenke, 2003). Anxiety Disorder. GAD-2 (Kroenke, 2007). Pittsburgh Sleep Quality Index (Buysse, 1989). Fatigue visual analogue scale. Fatigue Severity Scale (Krupp, 1989). Pain visual analogue scale. If diagnosed: Fibromyalgia Impact Questionnaire-R (Williams & Arnold, 2011); Roland-Morris Disability Questionnaire (Roland & Morris, 1983); PHQ 9 (Kroenke et al 2002); GAD 7 (Spitzer et al, 2006). Demographics (Baseline). Expectations for care (Baseline). Patient satisfaction. 2-items from the CAHPS (AHRQ, 2012).
Clinical indicators and biomarkers | 3-, 6-, and 12-months
  Composite:
  Complete metabolic panel, hypoglycemic medication, full lipid panel (TC, HDL, fasting triglycerides), lipid medication, TSH/T4, HbA1c, systolic and diastolic blood pressure, hypertension medication, BMI (height & weight), waist circumference, body fat composition, smoking status, cardiovascular disease risk (general and events), metabolic syndrome diagnosis.
Service Utilization Data and Health Insurance Claims Data | 3-, 6-, and 12-months; biennially

OTHER OUTCOMES:
Patient Experiences (Fidelity) | Monthly for the first 6 mos., then each 3 months for the rest of the first year, then every 6 months.
  Composite:
  Dimensions assessed: access to care, whole person care, promotion of self-care and wellness, practitioner communication style, shared decision-making, trust in the practitioner, perceived practitioner empathy, perceived health partnership, and demographic information (CAHPS - AHRQ, 2012; ACES - Safran et al, 1998); CARE - Mercer, et al, 2004).
Provider Experiences (Fidelity) | Monthly for the first 6 months, then each 3 months for the rest of the first year, then every 6 months
  Composite:
  Team Climate Inventory Short Version (TCI - Anderson & West, 1995; Loo & Loewen, 2002). Additional items were derived from a study of integrative medicine team practice (Gaboury, et al, 2010). Items on integrative team collaboration, integrative treatment planning, personal development, and clinical skills development were developed for the study.
Medical records chart audit (Fidelity) | Monthly for the first 6 months, then each Monthly first 6 months then q. 3 months for the rest of the first year, then every 6 months
  Composite:
  Evidence of principles and best practices of integrative medicine: Whole person assessment and treatment; patient-practitioner health partnership; use of both conventional and CAM methods; health promotion and prevention interventions; use of natural and least invasive treatments where possible (support for body's innate healing capacity); patient personal care support team/team-based approach; extended visits/spending adequate time with patients; access to comprehensive, integrated, care.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Maizes, MD, Principal Investigator — University of Arizona Arizona Center for Integrative Medicine; Sally E Dodds, PhD, Study Director — University of Arizona Arizona Center for Integrative Medicine
Locations (1):
- University of Arizona Integrative Health Center (UAIHC), Phoenix, Arizona, United States

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kroenke, K., Spitzer R.L. (2002). The PHQ-9: A new depression and diagnostic severity measure. Psychiatric Annals, 32, 509-521.
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Littman AJ, White E, Satia JA, Bowen DJ, Kristal AR. Reliability and validity of 2 single-item measures of psychosocial stress. Epidemiology. 2006 Jul;17(4):398-403. doi: 10.1097/01.ede.0000219721.89552.51. PMID 16641618
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Williams DA, Arnold LM. Measures of fibromyalgia: Fibromyalgia Impact Questionnaire (FIQ), Brief Pain Inventory (BPI), Multidimensional Fatigue Inventory (MFI-20), Medical Outcomes Study (MOS) Sleep Scale, and Multiple Ability Self-Report Questionnaire (MASQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S86-97. doi: 10.1002/acr.20531. No abstract available. PMID 22588773
- [Background] Roland M, Morris R. A study of the natural history of low-back pain. Part II: development of guidelines for trials of treatment in primary care. Spine (Phila Pa 1976). 1983 Mar;8(2):145-50. doi: 10.1097/00007632-198303000-00005. PMID 6222487
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Safran DG, Kosinski M, Tarlov AR, Rogers WH, Taira DH, Lieberman N, Ware JE. The Primary Care Assessment Survey: tests of data quality and measurement performance. Med Care. 1998 May;36(5):728-39. doi: 10.1097/00005650-199805000-00012. PMID 9596063
- [Background] Mercer SW, Maxwell M, Heaney D, Watt GC. The consultation and relational empathy (CARE) measure: development and preliminary validation and reliability of an empathy-based consultation process measure. Fam Pract. 2004 Dec;21(6):699-705. doi: 10.1093/fampra/cmh621. Epub 2004 Nov 4. PMID 15528286
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Loo, R & Loewen, P. (2002). A Confirmatory Factor-Analytic and Psychometric Examination of the Team Climate Inventory : Full and Short Versions. Small Group Research, 33: 254.
- [Background] Agency for Healthcare Research and Quality. (2012). Consumer Assessment of Healthcare Providers and Systems surveys. Accessed October 12, 2012 from the World Wide Web ar http://cahps.ahrq.gov/clinician_group.
- [Background] Gaboury I, Boon H, Verhoef M, Bujold M, Lapierre LM, Moher D. Practitioners' validation of framework of team-oriented practice models in integrative health care: a mixed methods study. BMC Health Serv Res. 2010 Oct 14;10:289. doi: 10.1186/1472-6963-10-289. PMID 20942973
- [Background] Bech P, Olsen LR, Kjoller M, Rasmussen NK. Measuring well-being rather than the absence of distress symptoms: a comparison of the SF-36 Mental Health subscale and the WHO-Five Well-Being Scale. Int J Methods Psychiatr Res. 2003;12(2):85-91. doi: 10.1002/mpr.145. PMID 12830302
- [Background] Centers for Disease Control and Prevention (2012). Behavioral Risk Factor Surveillance System Survey Questionnaire. Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention. Accessed October 15, 2012 from the World Wide Web at http://www.cdc.gov/brfss.
- [Background] Anderson, N. R., & West, M. A. (1998). Measuring climate for work group innovation: Development and validation of the team climate inventory. Journal of Organizational Behavior, 19, 235-258.
- [Derived] Herman PM, Dodds SE, Logue MD, Abraham I, Rehfeld RA, Grizzle AJ, Urbine TF, Horwitz R, Crocker RL, Maizes VH. IMPACT--Integrative Medicine PrimAry Care Trial: protocol for a comparative effectiveness study of the clinical and cost outcomes of an integrative primary care clinic model. BMC Complement Altern Med. 2014 Apr 7;14:132. doi: 10.1186/1472-6882-14-132. PMID 24708726